CLINICAL TRIAL: NCT00299013
Title: A Multicentre, Randomised, Double Blind, Double Dummy, Active Comparator Controlled, Parallel Group Study of COLAL-PRED® in the Treatment of Moderate Acute Ulcerative Colitis
Brief Title: Study of COLAL-PRED® in the Treatment of Moderate Acute Ulcerative Colitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Alizyme (Industry)
Responsible Party: Research and Development Director, Alizyme
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ATL2502/020/CL
Record Dates: First submitted 2006-03-02; First posted 2006-03-06 (Estimated); Last update posted 2008-04-25 (Estimated); Status verified 2008-04

CONDITIONS: Ulcerative Colitis
Keywords: Ulcerative colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Methylprednisolone; Prednisolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): Prednisolone 40mg oral tablets, once daily, dose tapering weekly (40,40,30,20,15,10,5,0mg) over 8 weeks.
  Interventions: Drug: Prednisolone
- 2 (Experimental): COLAL-PRED 40mg oral capsule, once daily for 8 weeks.
  Interventions: Drug: COLAL-PRED®
- 3 (Experimental): COLAL-PRED 60mg oral capsule, once daily for 8 weeks.
  Interventions: Drug: COLAL-PRED®
- 4 (Experimental): COLAL-PRED 80mg oral capsule, once daily for 8 weeks.
  Interventions: Drug: COLAL-PRED®

INTERVENTIONS:
Drug: COLAL-PRED® — COLAL-PRED 40, 60 or 80mg oral capsule, once daily for 8 weeks.
  Other Names: Prednisolone sodium metasulfobenzoate.
  Arms: 2; 3; 4
Drug: Prednisolone — Prednisolone 40mg oral tablets, once daily, dose tapering weekly (40,40,30,20,15,10,5,0mg) over 8 weeks.
  Arms: 1

SUMMARY:
The purpose of this study is to investigate whether a novel dosage form of a prednisolone ester, called COLAL-PRED®, is useful in the treatment of ulcerative colitis.

DETAILED DESCRIPTION:
Ulcerative colitis is a disease that causes inflammation of the large bowel, causing fever, diarrhoea, dehydration and other symptoms. Standard treatment for ulcerative colitis includes general medical treatments such as fluid and salt replacement and attention to diet. Anti-inflammatory medicines such as steroids (e.g. prednisolone) and aminosalicylates (e.g. mesalazine) are the main drug treatments.

This study will investigate whether COLAL-PRED®, a novel dosage form of a prednisolone ester, is safe and effective in the treatment of ulcerative colitis, compared with the standard treatment (conventional prednisolone) and also to determine which dose which will work best for future patients.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopically confirmed diagnosis of ulcerative colitis
* Score of 6-10 on the Disease Activity Index (DAI)
* Moderate to severe mucosal appearance

Exclusion Criteria:

* Previous colonic surgery
* Other treatments for ulcerative colitis that have not been stabilised
* Clinically significant diabetes, heart failure, unstable angina, cirrhosis, renal failure
* History of tuberculosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 796 (Actual)
Dates: Start 2006-03; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

PRIMARY OUTCOMES:
Disease activity index | After 4 and 8 weeks of treatment
Cortisol levels | After 4 and 8 weeks of treatment

SECONDARY OUTCOMES:
Simple clinical colitis activity index | 8 weeks
Endoscopy | 8 weeks
Adverse events | 12 weeks
Laboratory tests | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hawkey, Principal Investigator — University Hospital, Nottingham
Locations (86):
- Australia (3):
  - Research Site, Bankstown, New South Wales
  - Research Site, Bedford Park, South Australia
  - Research Site, Parkville, Victoria
- Belgium (3):
  - Research Site, Brussels
  - Research Site, Ghent
  - Research Site, Roeselare
- Czechia (11):
  - Gastroenterologicka ambulance, Hradec Králové
  - Hepato-Gastroenterologie HK s.r.o., Hradec Králové
  - Krajska nemocnice Liberec, Liberec
  - Research Site, Olomouc
  - Research Site, Prague
  - Privatni odborna ambulance, Prague
  - Oblastni nemocnice Pribram a.s., Příbram
  - Okresni nemocnice Tabor, Tábor
  - Nemocnice v Usti nad Orlici, Ústí nad Orlicí
  - Research Site, Zlín
  - Krajska nemocnice T Bati a s, Zlín
- Denmark (4):
  - Aalborg Hospital, Aalborg
  - Helsingors Hospital, Elsinore
  - Gentofte Hospital, Hellerup
  - Hvidovre Hospital, Hvidovre
- France (4):
  - CHU Nord Hepato-Gastroenterologie, Amiens
  - Hopital de l'Archet II, Nice
  - Hopital Saint Louis, Paris
  - Hospital Haut Leveque, Pessac
- Am Wallgraben 99, Stuttgart, Germany
- Hungary (11):
  - Research Site, Debrecen
  - Research Site, Dunaújváros
  - Research Site, Eger
  - Petz Aladar Megyei Korhaz, Győr
  - Bekes Megyei Kepviselotestulet Pandy Kalman Korhaza, Gyula
  - Research Site, Hatvan
  - Miskolc MJV Semmelweis Korhaz, Miskolc
  - Research Site, Szekszárd
  - Fejer Megyei Szent Gyorgy Korhaz, Székesfehérvár
  - Vas Megyei Markusovszky Korhaz, Szombathely
  - Research Site, Vác
- Israel (6):
  - Research Site, Haifa
  - Research Site, Jerusalem
  - Research Site, Kfar Saba
  - Research Site, Petah Tikva
  - Research Site, Rehovot
  - Research Site, Tel Aviv
- Policlinico S. Orsola-Malpighi, Bologna, Italy
- Poland (10):
  - Samodzielny Publiczny Szpital Kliniczny, Klinika Gastroenterologii i Chorob Wewnetrznych, Bialystok
  - SP ZOZ Uniwersytecki Szpital Kliniczny Nr 5 im. gen. dyw. Boleslawa Szareckiego Uniwersytetu Medycznego w Lodzi Oddział Gastroenterologii i Chorob Wewnetrznych, Lodz
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie Klinika Gastroenterologii, Lublin
  - Szpital Kolejowy w Pruszkowie Oddzial Wewnetrzny, Pruszków
  - SPSK Nr 1 im. Prof. Tadeusza Sokolowskiego Pomorskiej Akademii Medycznej Klinika Gastroenterologii i Chorob Wewnetrznych, Szczecin
  - Research Site, Torun
  - Research Site, Warsaw
  - Centrum Onkologii-Instytutu im. Marii Skłodowskiej-Curie Klinika Gastroenterologii, Warsaw
  - Samodzielny Publiczny Centralny Szpital Kliniczny w Warszawie Katedra i Klinika Gastroenterologii i Chorób Przemiany Materii, Warsaw
  - Wojskowy Szpital Kliniczny z Poliklinika Oddzial Gastroenterologii, Wroclaw
- Russia (2):
  - Research Site, Moscow
  - Research Site, Saint Petersburg
- South Africa (7):
  - Research Site, Port Elizabeth, Eastern Cape
  - Research Site, Cape Town, Western Cape
  - Kingsbury Hospital, Cape Town
  - Panorama Mediclinic, Cape Town
  - Parklands Medical Centre, Durban
  - Fordsburg Clinic, Johannesburg
  - Kloof Medi Clinic, Pretoria
- Spain (6):
  - Research Site, Córdoba, Andalusia
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario del Mar, Barcelona
  - Research Site, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario Joan XXIII, Tarragona
- Sweden (3):
  - Karolinska University Hospital Solna, Stockholm
  - Sophiahemmet Stockholm, Stockholm
  - Norrlands University Hospital Umea, Umeå
- United Kingdom (14):
  - Addenbrooke's Hospital, Cambridge
  - Research Site, Cottingham
  - Darent Valley Hospital, Dartford
  - Research Site, Edinburgh
  - Western General Hospital, Edinburgh
  - Leeds General Infirmary, Leeds
  - Leicester General Hospital, Leicester
  - Research Site, Liverpool
  - Hammersmith Hospital, London
  - Middlesex Hospital, London
  - Royal Victoria Infirmary, Newcastle upon Tyne
  - University Hospital, Nottingham
  - Hope Hospital, Salford
  - Research Site, Sheffield